CLINICAL TRIAL: NCT06836375
Title: Estudio Piloto Para la aplicación de Dispositivos bioelectrónicos Externos de Baja Potencia en el diagnóstico de Asma Bronquial
Brief Title: Pilot Study for the Application of Low Power External Bioelectronic Devices in the Diagnosis of Bronchial Asthma.
Status: Not yet recruiting | Type: Observational
Sponsor: Acurable Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1914-N-22
Record Dates: First submitted 2025-02-13; First posted 2025-02-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-02

CONDITIONS: Asthma Bronchiale
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Bronchial asthma: Patients with a diagnosis of bronchial asthma, under follow-up by the Asthma Unit.
  Interventions: Diagnostic Test: Spirometry test with bronchodilation; Diagnostic Test: Methacholine challenge; Diagnostic Test: impulse oscillometry; Other: Measurement of the exhaled FeNO fraction
- Patients referred for consultation: Patients referred for consultation due to clinical suspicion of bronchial asthma.
  Interventions: Diagnostic Test: Spirometry test with bronchodilation; Diagnostic Test: Methacholine challenge; Diagnostic Test: impulse oscillometry; Other: Measurement of the exhaled FeNO fraction

INTERVENTIONS:
Diagnostic Test: Spirometry test with bronchodilation — this test measures how much air you can breathe in and out of your lungs, as well as how easily and fast you can then blow the air out of your lungs
Diagnostic Test: Methacholine challenge — test used to diagnose asthma where the patient breaths in methacholine
Diagnostic Test: impulse oscillometry — test that uses sound waves to measure how much resistance there is to the normal movement of air in and out of your lungs when you are breathing at rest
Other: Measurement of the exhaled FeNO fraction — Measure the level of nitric oxide in parts per billion (PPB) in the air the patient slowly exhales

SUMMARY:
The objective of this study is to detect the acoustic signals generated by the respiratory system on asthma patients using an acoustic sensor and retrospectively use these signals to identify the characteristics that differentiate patients with asthma and healthy subjects.

DETAILED DESCRIPTION:
The objective of this project is to detect acoustic signals generated by the respiratory system in patients with asthma using the acoustic sensor; and then, retrospectively, to use these signals to carry out signal processing research, with the aim of trying to identify signal characteristics that can be used to differentiate asthma patients from people who do not have the disease.

The hypothesis, therefore, is that it is possible to target through external smart bioelectronic devices and wireless connectivity (wearables) the initial signals of the pathophysiology of bronchial asthma and differentiate them from the signals of the normal respiratory physiology of a healthy individual.

Similarly, detection of such signals would not only be useful for asthma diagnosis but also for monitoring and early detection of exacerbations before they can be detected by the usual respiratory functional tests.

The patients will first visit the asthma unit where the diagnostic tests will be undertaken. Then the subjects will take the acoustic sensor home with them and wear it during sleep for at least two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged >= 18 and < 65.
* Ability to access applications on mobile device, technical understanding and minimal technological skills
* Subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

* Subject does not consent to the study
* Subject does not comply with inclusion criteria
* Subject has a known allergy to medical adhesives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from or referred to the asthma unit in the hospital Virgen del Rocio in Seville, Spain
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-27 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2027-02-27 (Estimated)

PRIMARY OUTCOMES:
Acoustic respiratory signals | During the diagnostic tests performed and during the night studies performed by the participant for at least two weeks
  Acoustic signals during the tests performed for asthma diagnosis and while the subjects sleep for at least two weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Virgen del Rocio, Seville, Spain

IPD SHARING:
Plan to Share IPD: No